CLINICAL TRIAL: NCT07015593
Title: Patient Journey in Conventional Therapy for Primarily Treated Advanced Gynecologic Cancers in China
Brief Title: Patient Journey in Advanced Gynecologic Cancers
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Gang Chen (101199), Prof, Tongji Hospital
Other Study IDs: NIS103233; [2024]S257 (Other: Medical Ethics Committee of Tongji Medical College, HUST)
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Genital Neoplasms, Female; Uterine Cervical Neoplasms; Endometrial Carcinoma
MeSH Terms: conditions — Genital Neoplasms, Female; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: 780 patients for interview
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — 30 for Qualitative interview and 750 for quantitative survey

SUMMARY:
This is a mixed-methods survey study including a 2-phased sequential-explanatory design. This study is to understand the patient journey in conventional therapy for newly diagnosed stage III or IV CC or EC in China, including ①patients' treatment decision making factors and treatment experiences and ② patients' unmet needs during post-treatment surveillance.

DETAILED DESCRIPTION:
This is a mixed-methods survey study including a 2-phased sequential-explanatory design: Phase 1, Qualitative interview will be done first to explore the treatment decision factors, treatment experiences and unmet needs during post treatment surveillance, to provide components and inform the quantitative data collection. Phase 2, quantitative survey to collect data on a larger scale and allow a statistical generation of the qualitative findings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Newly diagnosed stage III or IV CC or EC
* Completed their initial conventional therapies which must include at least chemotherapy, radiotherapy or a combination between Dec. 2022 to Dec. 2024 and the therapies were within 6 months after diagnosis.
* Told by their physician that their disease is stable.
* Patients must have informed consent form (ICF) signed for the study.

Exclusion Criteria:

* Previously treated with targeted biologic therapy anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
* Previously participated in or participating in a clinical trial.
* Patients who received another line of therapy after initial therapy.
* Unable or unwilling to provide informed consent.
* Not fluent in local language.
* Indicates or exhibits hearing difficulties, which would make a conversation challenging.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is estimated that ~780 patients will be included in this study. For qualitative insights, previous studies have shown that a minimum of 12 respondents (Guest et al. 2006) is required to reach data saturation. A sample size of ~30 will be sufficient to gather qualitative insights and attain saturation. For quantitative survey, considering most of the variables in quantitative survey are categorical variables, we tend to use 50% in the sample size formula since it will provide us with the maximum sample size required for any question, we calculated the sample size to be ~750 with a confidence interval of 95% and margin of error 5%. The number of specific experts interviewed may be fine-tuned depending on actual implementation.
Sampling Method: Non-Probability Sample
Enrollment: 780 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Treatment decision making | 1 day. At the time of the interview.
  1. Information seeking in treatment decision
  2. Treatment decision making factors
  3. Clinical trial awareness
Initial treatment experiences | 1 day. At the time of the interview.
  1. Influence of treatment on daily life and work
  2. Information and education during treatment
  3. Coordination of care
  4. Overall impression on care received and doctor/nurses' availability
Unmet needs and gaps from diagnosis to post-treatment surveillance | 1 day. At the time of the interview.
  1. Psychological and emotional needs
  2. Social support needs
  3. Healthcare needs
  4. Gaps during follow-up care

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, PhD, Principal Investigator — Tongji Hospital
Locations (4):
- China (4):
  - Ying Zhou, Hefei, Anhui
  - Shuzhong Yao, Guangzhou, Guangdong
  - Gang Chen, Wuhan, Hubei
  - Dongling Zou, Chongqing

IPD SHARING:
Plan to Share IPD: No